CLINICAL TRIAL: NCT00838955
Title: Temsirolimus for Relapsed/Refractory Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: There was lack of enrollment since January 2013
Sponsor: Loyola University (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Hagen, Patrick A, Associate Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201170
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin's lymphoma; relapsed Hodgkin's lymphoma; refractory Hodgkin's lymphoma; Temsirolimus
MeSH Terms: conditions — Hodgkin Disease | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temsirolimus (Experimental): Temsirolimus 25 mg IV infusion on Days 1, 8, 15, and 22 of a 28 day cycle
  Interventions: Drug: Temsirolimus

INTERVENTIONS:
Drug: Temsirolimus — Temsirolimus 25 mg IV infusion on Days 1, 8, 15, and 22 of a 28 day cycle

SUMMARY:
This clinical trial is for patients with Hodgkin Lymphoma that has not responded to standard treatment. The purpose of this study is to determine what effects, good or bad, Temsirolimus has on Hodgkin Lymphoma. The study will also determine whether Temsirolimus is tolerated in patients with Hodgkin Lymphoma who have been previously treated with chemotherapy.

DETAILED DESCRIPTION:
Temsirolimus 25 mg IV infusion will be given once weekly on days 1, 8, 15 and 22 of each cycle. Patients will be assessed for response with CT scans after the second cycle, and then after every other cycle until disease progression is confirmed.

Patients will be treated with Temsirolimus until disease progression, or up to six cycles. Continuation of therapy beyond cycles is at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed classical Hodgkin Lymphoma or Lymphocyte Predominant Hodgkin Lymphoma with progressive disease during or at the end of the previous therapy, as defined by the IWG criteria.
* Patient must have nodular sclerosing, lymphocyte depleted, or mixed cellularity Hodgkin Lymphoma (Classical Hodgkin Lymphoma), or Lymphocyte predominant Hodgkin Lymphoma.
* Baseline measurements and evaluations must be obtained within 4 weeks of registration to the study.
* Abnormal PET scans will not constitute evaluable disease, unless verified by CT scan or other appropriate imaging.
* A clearly defined, bidimensionally measurable lymph node or tumor mass measuring at least 2 cm in diameter on a CT scan.
* Patient should have had at least one line of prior chemotherapy. Patients relapsing after treatment with radiation therapy alone are not eligible.
* Age > than or equal to 18 years.
* Both men and women and members of all races and ethnic groups are eligible for this trial.
* Women must not be pregnant or breast-feeding due to lack of information about the safety of administration of Temsirolimus in pregnant and lactating patients. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy.
* Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of pregnancy prevention.
* Patient must have a SWOG performance status between 0-2.
* Patient must have no prior treatment with an m-TOR inhibitor.
* Patient must not have active infections at the time of registration.
* Laboratory studies should be obtained within two weeks of study registration except where noted otherwise. Allowable laboratory values are listed below:
* Absolute neutrophil count > than or equal 1,000/mm3
* Hemoglobin > than or equal 8 gm/dL
* Platelets > than or equal 75,000/mm3
* Serum creatinine < than or equal to two times the upper limit of normal. Creatinine should be measured within seven days of registration.
* Total serum bilirubin < than or equal to ≤ 1.5 times the upper limit of normal. Total bilirubin should be measured within seven days of registration.
* AST (SGOT) < than or equal to 3 times the upper limit of normal.
* ALT (SGPT) < than or equal to 3 times the upper limit of normal.
* Fasting total cholesterol < than or equal to 350 mg/dL.
* Fasting triglyceride level < than or equal to 400 mg/dL.
* Patient must have a life expectancy of three months.

Exclusion Criteria:

* Patient must not have received prior allogeneic stem cell transplantation. Prior autologous stem cell transplantation more than six months prior to registration is acceptable.
* Patient must not have received prior chemotherapy, biologic therapy or radiation within three weeks prior to registration, and should have recovered from toxicities of prior therapy (to Grade 0 or 1).
* Patient must not have evidence of active CNS disease.
* Patient must not have an uncontrolled comorbid disease, including hyperlipidemia, hypertriglyceridemia, diabetes mellitus, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Patient must not have a psychiatric illness or social situation that would limit compliance with study requirements.
* Patient must have a life expectancy of three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-01; Primary Completion 2016-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
To estimate the overall response rate (complete or partial response and stable disease by the IWG criteria) to temsirolimus | 26 weeks
  To estimate the overall response rate (complete or partial response and stable disease by the IWG criteria) to temsirolimus

SECONDARY OUTCOMES:
To evaluate the toxicity of temsirolimus in this patient population. | 26 weeks
  To evaluate the toxicity of temsirolimus in this patient population.
To estimate the time to progression after treatment with temsirolimus. | 5 years
  To estimate the time to progression after treatment with temsirolimus.
To estimate overall survival after treatment with temsirolimus. | 5 years
  To estimate overall survival after treatment with temsirolimus.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Hagen, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola Univeristy Medical Center, Cardinal Bernardin Cancer Center, Maywood, Illinois, United States